CLINICAL TRIAL: NCT06544356
Title: The Effect of Mothers' Health Literacy Levels on Their Knowledge and Attitudes Towards Newborn Screenings
Brief Title: Health Literacy and Newborn Screenings
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Abdullah Adiyaman, Graduate Student, Yuzuncu Yil University
Other Study IDs: YuzuncıYıl 2
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Health Literacy and Newborn Screening
Keywords: health literacy; newborn screening programme; mother; newborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One grups: Mums who've just given birth, Over 18 years of age, literate mothers with at least primary school education
  Interventions: Other: No intervention, questionnaire filled out

INTERVENTIONS:
Other: No intervention, questionnaire filled out — Mother introductory information form, Health Literacy Scale, Knowledge and Attitude Scale about Newborn Screenings were completed.

SUMMARY:
Health literacy, the ability to understand and use health information, is crucial in all health processes such as healthy living, disease prevention, diagnosis, treatment, and personal care. The newborn screening program (NSP) helps reduce morbidity and mortality by early diagnosing rare diseases in infants. Health literacy impacts parents' vaccination choices and attitudes, and higher health literacy is sometimes associated with lower adherence to vaccination protocols. Various studies highlight the significance of health literacy in childhood vaccinations, breastfeeding effectiveness, and attitudes toward YTP, emphasizing parents' lack of knowledge about NSP and the need for education. Notably, parents who give birth outside of hospitals have significant knowledge gaps regarding NSP.

DETAILED DESCRIPTION:
Health literacy involves clearly communicating and accurately understanding health information. It is defined as being related to all points in the care process, from promoting and enhancing healthy living to preventing and detecting diseases, diagnosing and decision-making, treating, and personal care.

The newborn screening program (YTP) is defined as the early diagnosis of rare presymptomatic congenital diseases by analyzing blood samples taken from infants' heels. YTP has been stated to significantly reduce morbidity and mortality rates in infants. YTP is used to detect many diseases, including hearing loss, congenital heart defects, endocrine disorders, hemoglobinopathies, congenital metabolic diseases, cystic fibrosis, spinal muscular atrophy, lysosomal storage disorders, and immunodeficiencies.

One study found that communicative health literacy was directly related to vaccination adherence compared to functional and critical health literacy. Parents with higher levels of communicative and critical health literacy were less likely to fully adhere to vaccination protocols. Attitudes towards vaccines and beliefs about the reliability of unofficial vaccine information sources serve as directly related factors in vaccination practices and are reported to mediate the relationship between health literacy and vaccination adherence.

Another study showed that health literacy was related to parents' preferences for the rotavirus vaccine. When vaccines were offered in the free market, parents with higher health literacy were less likely to vaccinate their newborns against rotavirus compared to parents with lower health literacy.

A descriptive study conducted with 279 parents of children aged 0-12 months in the central district of Kırıkkale province found that health literacy was not related to attitudes and behaviors towards childhood vaccinations.

In a study with a Latino population, one-third were found to have inadequate health literacy when measured by reading comprehension, and eight out of ten were inadequate when measured primarily by arithmetic. Furthermore, a significant relationship was reported between limited health literacy levels and lower antibiotic knowledge among Latino parents.

A study found that mothers' health literacy levels and breastfeeding effectiveness were adequate before hospital discharge. The study also indicated that health literacy level served as a protective factor against stopping breastfeeding.

Another study found that most mothers lacked knowledge about blood spots. Additionally, mothers believed that researching dried blood spots was a good thing.

A study evaluating mothers' views on YTP reported that 51.4% of mothers found their knowledge about newborn screening tests partially sufficient and 66.3% wanted information from healthcare personnel. It was also found that 54.8% of mothers knew some diseases could be inherited, 56% knew that genetic diseases were caused by consanguineous marriage, 51.3% knew these diseases could cause irreversible brain damage in infants, 42% knew they could lead to physical growth and development delays, and 48% knew that a diagnosis could be made with two drops of blood taken from the baby's heel. The study emphasized the important roles that nurses and other healthcare professionals should play.

A study evaluating the knowledge and attitudes of midwives and parents who gave birth outside hospitals regarding YTP indicated that midwives informed parents who gave birth in hospitals about YTP. However, parents who gave birth outside hospitals had significant knowledge gaps about YTP and expressed a desire for education on the subject

A study assessing various experiences and attitudes towards YTP found that while parents generally had a positive view of the screening process, some participants experienced significant frustration, particularly regarding how results were received.

ELIGIBILITY:
Inclusion Criteria:

* Newly delivered mothers,
* At least primary school graduate and literate,
* Over 18 years of age,
* Accepted voluntary participation in the research,
* Mothers open to communication.

Exclusion Criteria:

* Single individuals or without children,
* Under 18 years of age,
* Illiterate,
* Who did not accept voluntary participation in the research,
* Mums out of touch.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Mothers who gave birth in the hospital, were hospitalised in puerperal wards and met the study criteria.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Health Literacy Scale | 6 monts
  The Health Literacy Scale (HLS-14) was used. The scale consists of three sub-dimensions: Functional Health Literacy (5 items), Interactive Health Literacy (5 items), and Critical Health Literacy (4 items). The scale has a maximum score of 70 and a minimum score of 15. The higher the score, the higher the level of health literacy.

SECONDARY OUTCOMES:
Knowledge and Attitude Scale about Newborn Screening | 6 monts
  The Knowledge and Attitude Scale Regarding Newborn Screenings, adapted into was used. The scale has a maximum score of 52 and a minimum score of 0. The higher the score, the lower the level of knowledge and attitudes about newborn screening.

OTHER OUTCOMES:
Maternal Introductory Information Form | 6 monts
  For the determination of socio-demographic characteristics, the 24-question Maternal Introductory Information Form, which was prepared by using the literature, was used.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Adıyaman, Principal Investigator — abdullah.adiyaman@erzurum.edu.tr
Locations (1):
- Van Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No